CLINICAL TRIAL: NCT03145220
Title: Randomized Double Blind Placebo-controlled Phase II Study on the Effects of EA-230 on the Systemic Inflammatory Response Following On-pump Cardiac Surgery
Brief Title: Immunomodulation of EA-230 Following On-pump Coronary Artery Bypass Grafting (CABG)
Acronym: EASI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Exponential Biotherapies Inc. (Industry)
Responsible Party: Principal Investigator, Peter Pickkers, prof. dr., Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EASI-Study; 2015-005600-28 (EudraCT Number)
Record Dates: First submitted 2016-06-22; First posted 2017-05-09 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Systemic Inflammatory Response Syndrome; Coronary Artery Bypass Grafting
Keywords: EA-230; Systemic Inflammatory Response Syndrome; Acute Kidney Injury; Interleukin-6; Safety; Tolerability; Phase II; Randomized clinical trial
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Acute Kidney Injury | interventions — alanyl-glutaminyl-glycyl-valine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EA-230 (Active Comparator): Intravenous infusion of EA-230, 90 mg/kg/hour. Administered from start of surgical incision until stoppage of the cardio-pulmonary bypass pump, for a maximum of 4 hours.
  Interventions: Drug: EA-230
- Placebo (Placebo Comparator): Intravenous infusion of NaCl (equivalent osmolarity with active intervention EA-230). Administered from start of surgical incision until stoppage of the cardio-pulmonary bypass pump, for a maximum of 4 hours.
  Interventions: Other: Placebo (NaCl)

INTERVENTIONS:
Drug: EA-230 — Active intervention
  Other Names: AQGV
  Arms: EA-230
Other: Placebo (NaCl) — Placebo intervention
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
EA-230 is a newly developed synthetic compound with anti-inflammatory properties, it is a linear tetrapeptide derived from the human chorionic gonadotropin hormone (hCG). Recently, its immunomodulatory effects in humans were confirmed in a phase I trial and an optimal dose was established. To establish this anti-inflammatory effect in a selected patient population and assess clinical outcome, a combined phase IIa/IIb trial will be conducted with patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Systemic inflammation is a condition in which the innate immune system is activated due to a variety of causes such as sepsis, trauma, and major surgical interventions. The clinical condition in which the body responds to such stimuli by the release of circulating inflammatory mediators is well known as the systemic inflammatory response syndrome (SIRS) and is defined by tachypnoea, tachycardia, leucocytosis or leucopenia and hyper- or hypothermia.

Although this activation of the immune system is essential for survival, the often subsequent overwhelming pro-inflammatory response may be detrimental. Of the many downstream consequences of this exaggerated inflammatory response, organ injury and failure is the most serious, most often involving the kidneys. Multiple organ failure (MOF) is associated with high morbidity and mortality, whereas failure of kidneys is an independent prognostic factor for mortality in critically ill patients.

This exaggerated systemic pro-inflammation also occurs during major surgical procedures, especially in cardiac surgery procedures. Multiple stimuli during these procedures, such as sternotomy, extra-corporal cardio-pulmonary bypass (ECC) and aortal cross-clamping, account for substantial systemic inflammatory activation. The extent of inflammation following this procedures is directly associated with patient outcome, as high post-operative levels of IL-6 have been proven to correlate with adverse outcome and mortality. Also at organ level, the incidence of inflammation associated development of acute kidney injury (AKI) following cardiac surgery is high and correlates with adverse outcome and mortality.

To date, no immunomodulatory treatments, aimed at dampening the (acute) systemic inflammatory reaction following cardiac surgery with cardio-pulmonary bypass, have shown to improve essential outcome. Current strategies consist of prevention and supportive treatment; new strategies aiming at attenuating this exaggerated pro-inflammatory response are therefore warranted.

EA-230 is a novel pharmacological compound, developed for the treatment of systemic inflammation and associated organ dysfunction. It is a linear tetrapeptide derived from the human chorionic gonadotropin hormone (hCG). It has shown anti-inflammatory properties and protects against organ failure and associated mortality in several pre-clinical models of sepsis or systemic inflammation. As EA-230 attenuates the pro-inflammatory response in neutrophils and monocytes ex vivo, and neutrophil influx in tissues during systemic inflammation in vivo is abrogated, it is thought that EA-230 acts by protecting the host against the detrimental effects of neutrophils during acute systemic inflammatory diseases, thereby preventing organ damage.

A recently performed phase I study into the safety and tolerability of EA-230 in 24 subjects showed that continuous administration of EA-230 up to 90 mg/kg/hour infused intravenously is well tolerated and has an excellent safety profile. This profile was confirmed in a consequent executed phase IIa study in which 36 healthy subjects received the same dosages of EA-230 during human experimental endotoxemia. In this human model of controlled systemic inflammation elicited by the administration of a low dose of endotoxin, the anti-inflammatory effects of EA-230 shown in pre-clinical studies were confirmed and the optimal dose was established. Subjects treated with the highest dose (90 mg/kg/hour) showed less flu-like symptoms, development of fever was suppressed, and reduced levels of pro-inflammatory mediators (among others Interleukin-6 and Interleukin-8) were observed compared to placebo-treated subjects.

This current study is a combined phase IIa/IIb, randomized, placebo-controlled, double-blind, clinical trial. In the first part, phase IIa, the study aims to confirm safety and tolerability in a patient population (n=60, 30 active and 30 placebo) with systemic inflammation elicited by on-pump cardiac surgery. In the second part, phase IIb, the immunomodulatory effect of EA-230 is studied in a same patient population (n=180, 90 active and 90 placebo, including patients from part 1).

After inclusion of 90 patients, halfway the study, an additional adaptive power analysis will be performed to re-evaluate group size and power. Efficacy and sample size re-determination will be performed by the statistician of the Data Safety Management Board (DSMB).

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for elective on-pump CABG surgery.

   * Part 1: 60 patients undergoing CABG surgery, of which circa 40 low risk patients without valve replacement (range: 35-45)
   * Part 2: CABG surgery with or without valve replacement
2. Written informed consent to participate in this trial prior to any study-mandated procedure.
3. Patients aged >18, both male and female.
4. Patients have to agree to use a reliable way of contraception with their partners from study entry until 3 months after study drug administration.

Exclusion Criteria:

1. Immunocompromised

   * Solid organ transplantation
   * Known HIV
   * Pregnancy
   * Systemic use of immunosuppressive drugs
2. Non-elective/Emergency surgery
3. Hematological disorders

   * Known disorders from myeloid and/or lymphoid origin
   * Leucopenia (leucocyte count < 4x109/L)
4. Known hypersensitivity to any excipients of the drug formulations used
5. Treatment with investigational drugs or participation in any other intervention clinical trial within 30 days prior to study drug administration
6. Inability to personally provide written informed consent (e.g. for linguistic or mental reasons)
7. Known or suspected of not being able to comply with the trial protocol.

   In addition, for part 1 only (to select low-risk patients):
8. Euroscore II <4
9. Kidney function impairment: serum creatinine >200 µmol/L
10. Liver function impairment: Alanine transaminase/Aspartate transaminase (ALAT/ASAT) >3 times above upper level of reference range
11. Left ventricular dysfunction: Ejection fraction<35%
12. CABG procedure with valve replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-06; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability (treatment related (serious) adverse events) | Total (serious) adverse events related to treatment at day 90 after treatment
  Safety and tolerability expressed in treatment related (serious) adverse events
Interleukin-6 (IL-6) | 1 day: at baseline, start of the cardiopulmonary bypass (CPB), stop of CPB, 2h after stop of CPB, 4h after stop of CPB, 6h after stop of CPB and first post-operative day.
  Blood plasma levels IL-6

SECONDARY OUTCOMES:
Glomerular filtration rate (GFR) | Up to 3 days. At the day before surgery (baseline) and at the morning of the first post-operative day
  GFR assessed by plasma clearance of Iohexol.
Urine kidney injury markers (KIM-1, NGAL, L-FABP, TIMP-2*IGFBP-7, urinary IL-18, NAG, creatine, urea, albumin) | Up to1 day: at baseline (before surgery), 2h after stop of CPB, 4h after stop of CPB, 6h after stop of CPB and first post-operative day.
  laboratory values
Other cytokines/chemokines (TNFα, IL-8, IL-10, IL-1RA, MCP-1, MIP1α, MIP1β, VCAM, ICAM, IL-17A) | Up to 1 day: at baseline, start of the cardiopulmonary bypass (CPB), stop of CPB, 2h after stop of CPB, 4h after stop of CPB, 6h after stop of CPB and first post-operative day.
  Laboratory values.
Leukocyte counts (differentiated) | Up to 1 day: at baseline, start of the cardiopulmonary bypass (CPB), stop of CPB, 2h after stop of CPB, 4h after stop of CPB, 6h after stop of CPB and first post-operative day.
  Plasma leukocyte response, quantified by change of total cell counts, differentiated in lymphocytes, neutrophils, monocytes, basophils and eosinophils.

OTHER OUTCOMES:
Heart rate | First 24 post-operative hours, mean values per 30 minutes.
  Rate in beats per minute
Blood pressure | First 24 post-operative hours, mean values per 30 minutes.
  Pressure in mmHg
body temperature | First 24 post-operative hours, measured with an interval of 2 hours.
  Changes in body temperature in °C over time.
SOFA score (Sepsis-related Organ Failure Assessment score) | First 24 post-operative hours, twice.
  Change in SOFA score
Insulin sensitivity | First 24 post-operative hours.
  According to insulin dosing and plasma glucose concentration
length of stay on ICU (LOS ICU) | Up to 90 days.
  LOS ICU defined by total amount of days and hours patient is admitted to the intensive care
length of hospital stay (LOS) | Up to 90 days
  LOS defined by total amount of days and hours patient is hospitalized.
mortality | at day 28 and day 90
  28 and 90-days mortality
Major clinical adverse events | up to 90 days
  Incidence of major clinical adverse events within 90-days (stroke, MI, rethoracotomy, readmission, pleural and/or pericardial punction
APACHE IV | 1 day
  APACHE IV score at ICU admission
Other GFR methods (ECC) | ECC: Urine collection from start of surgery until the morning of the first post-operative day.
  Calculated endogenous clearance of creatine (ECC)
Other GFR methods (MDRD) | Before surgery (baseline) and all other days creatine is measured during during hospital stay (max 7 days)
  Estimated GFR with plasma creatinine: MDRD.
Plasma kidney function markers | Up to 7 days: At baseline (before surgery), at stop of CPB, 2h after stop of CPB, 4h after stop of CPB, 6h after stop of CPB, 12h after stop of CPB, first post-operative day and at all other days creatine is measured during during hospital stay
  Plasma creatinine and proenkephalin
Urine output | 1 day
  Modulation by EA-230 of changes in urine output in mL
Urinary laboratory parameters | baseline pre-operative and post-operative until day +1
  Changes in urea, sodium, creatinine and albumin in urine over time
Renal replacement therapy (RRT) | up to 90 days
  Need for and length of RRT
AKI stages | up to 90 days
  incidence of different stages of AKI according to the RIFLE criteria.
Vasopressor use | up to 7 days. Every 2 hours in the first 24-hours. Then once a day.
  Vasopressor use expressed as inotropic score ((dopamine dose × 1 µg/kg/min) + (dobutamine dose × 1 µg/kg/min) + (adrenaline dose × 100 µg/kg/min) + (noradrenaline dose × 100 µg/kg/min) + (phenylephrine dose × 100 µg/kg/min)) and ratio of inotropic score to the mean arterial pressure (MAP)
Fluid Therapy | First 24 post-operative hours, registered every 6 hours.
  Fluid therapy within the first 24 hours post-op. Expressed in total fluids administered, urine production and drain production.
Fluid balance | 7 days
  net fluid balance measured once a day (morning)
Cardiac injury markers | First 24 post-operative hours, twice.
  Change in plasma CK (Creatine kinase) and Troponin-t.
Chest drain production | During ICU admission, until removal of drains
  Chest drain production measured in mL
Cardioplegia fluid | up to 4 hours
  Cardioplegia fluid used during surgery: blood or crystalloid
Time until detubation | up to 90 days
  Time until post-operative detubation, measured in hours
A-a O2 gradient | First 24 post-operative hours, twice.
  Change in A-a O2 gradient.
Pharmacokinetics (PK) of EA-230 (Cmax, t1/2, Clearance, volume of distribution) | up to 6 hours: Sampling times in minutes after stop of CPB: t=0 (stop CPB), 1, 2, 5, 10, 20, 30, 60, 120, 240, 360.
  Complete PK-profile (Cmax, t1/2, Clearance, volume of distribution) of EA-230, only for a limited amount of patients (n=15)
Peak plasma levels of EA-230 (Cmax) | up to 4 hours. At start of CPB and at stop of CPB.
  Plasma peak levels of EA-230

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive care, research unit, Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Groenendael R, Beunders R, Hemelaar P, Hofland J, Morshuis WJ, van der Hoeven JG, Gerretsen J, Wensvoort G, Kooistra EJ, Claassen WJ, Waanders D, Lamberts MGA, Buijsse LSE, Kox M, van Eijk LT, Pickkers P. Safety and Efficacy of Human Chorionic Gonadotropin Hormone-Derivative EA-230 in Cardiac Surgery Patients: A Randomized Double-Blind Placebo-Controlled Study. Crit Care Med. 2021 May 1;49(5):790-803. doi: 10.1097/CCM.0000000000004847. PMID 33591006
- [Derived] van Groenendael R, Beunders R, Hofland J, Morshuis WJ, Kox M, van Eijk LT, Pickkers P. The Safety, Tolerability, and Effects on the Systemic Inflammatory Response and Renal Function of the Human Chorionic Gonadotropin Hormone-Derivative EA-230 Following On-Pump Cardiac Surgery (The EASI Study): Protocol for a Randomized, Double-Blind, Placebo-Controlled Phase 2 Study. JMIR Res Protoc. 2019 Feb 6;8(2):e11441. doi: 10.2196/11441. PMID 30724734